CLINICAL TRIAL: NCT00103961
Title: Primary HIV & Early Disease Research: American Cohort (PHAEDRA) AIEDRP
Brief Title: An Observational Study of People Who Have Recently Been Infected With HIV
Status: Completed | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Suzane Bazner, NP, Partners Healthcare
Other Study IDs: 5U01AI052403 (NIH); 2003-P-001991; 5U01AI052403 (NIH)
Record Dates: First submitted 2005-02-17; First posted 2005-02-18 (Estimated); Last update posted 2018-11-28 (Actual); Status verified 2008-09

CONDITIONS: HIV Infections
Keywords: Acute Infection; HIV; AIDS; Acute HIV; Early HIV
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood collection

GROUPS / COHORTS (1):
- 1: Treatment-naive and treatment-experienced HIV-infected adults
  Interventions: Behavioral: Questionnaire

INTERVENTIONS:
Behavioral: Questionnaire — A behavioral questionnaire will occur at Week 8

SUMMARY:
This is a long-term follow-up study of people who are identified during acute or recent HIV infection and are being followed at clinical research sites associated with the Acute HIV Infection and Early Disease Research Program (AIEDRP). The purpose of this study is to collect data on the immunological and virologic responses that occur early in the course of HIV infection in treatment-naive and treatment-experienced HIV infected adults.

Study hypothesis: This study will examine the immunological responses that occur early in the course of HIV infection in treated and untreated individuals. The long-term follow-up of these subjects will help identify host immunological and genetic factors along with therapeutic strategies associated with control of viremia and delayed disease progression. In addition, this cohort will provide the recruiting mechanism to support future trials of therapy to restore immune function. Furthermore, this cohort will provide a population suitable to monitoring changing patterns in the transmission of drug resistant viral strains while also evaluating ongoing behavioral risk factors associated with HIV transmission.

DETAILED DESCRIPTION:
This study will collect data on the immunological and virologic responses that occur early in the course of HIV infection in treated and untreated HIV infected adults to identify host immunological, virological, and therapeutic factors that influence disease progression. This study will also monitor changing patterns in the transmission of drug-resistant viral strains and evaluate ongoing behavioral risk factors associated with HIV infection.

Participants in this study will be followed for up to 10 years. During the first year of participation, study visits will occur approximately every 4 weeks for the first 12 weeks, then every 12 weeks thereafter, with a minimum of 8 study visits during the first year. Participants will be asked to complete a behavioral questionnaire at Week 8. After the first year of participation, there will be 4 visits per year. Blood collection and vital sign measurement will occur at each study visit.

Participants enrolled in this study are strongly encouraged to also enroll in the AIEDRP CORE01 study.

ELIGIBILITY:
Inclusion Criteria:

* Documented acute or recent HIV infection as defined in the study protocol
* Willing to be followed longitudinally by this study

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Treatment-naive and treatment-experienced HIV-infected adults
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2004-01; Primary Completion 2007-10 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric Rosenberg, MD, Principal Investigator — Partners Healthcare, Massachusetts General Hospital; Bruce D. Walker, MD, Principal Investigator — Partners Healthcare, Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Brigham & Women's Hospital, Boston, Massachusetts

REFERENCES:
- See also: Click here for more information on AIEDRP CORE01 — http://clinicaltrials.gov/ct/show/NCT00086372